CLINICAL TRIAL: NCT02082171
Title: Multidomain Intervention to Prevent Disability in Elders
Acronym: MINDED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C12-55; 2013-A00380-45 (Registry Identifier: IDRCB)
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2021-08

CONDITIONS: Physical Frailty; Physical Disability; Mobility Disability
Keywords: older adults; physical disability; multidomain intervention; prevention; pilot study; frailty; mobility; comprehensive geriatric assessment
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (No Intervention)
- Intervention group (Experimental): Comprehensive geriatric assessment followed by multi-domain preventive intervention
  Interventions: Other: Multidomain intervention

INTERVENTIONS:
Other: Multidomain intervention — Multidomain preventive intervention designed by a multidisciplinary team on the basis of results of a comprehensive geriatric assessment
  Arms: Intervention group

SUMMARY:
Prevention of physical disability represents a major priority for the public health system. Physical disability is the final result of a complex cascade of negative events occurring at different levels (i.e., environmental, social, biological, and clinical). The heterogeneity of the underlying mechanisms responsible for the onset of physical disability may require the adoption of preventive interventions affecting multiple domains. Although several studies suggest that single or different combinations of preventive interventions (in particular, physical activity, cognitive training, and healthy diet) might provide beneficial effects in preventing functional loss (and its related features, such as pain or reduced quality of life), very limited evidence coming from clinical trials is currently available on the topic. Intervention trials are usually designed to test the effect of a specific monodimensional intervention on a very selected population, so to reduce the risk of biased results. This approach, although legitimate and methodologically correct, may 1) be insufficient to target the multiple and heterogeneous physiopathological mechanisms underlying the onset of physical disability, and 2) cause a population selection bias leading to difficulties in implementing the study results to the overall older population (thus, determining the "evidence-based medicine" issue in the elderly). To our knowledge, there are no available data from clinical trials evaluating the effects of a multidomain intervention based on lifestyle modifications (e.g., physical activity, cognitive training, nutritional modification) for preventing mobility disability (a very early phase of the disabling process) in community-dwelling older persons. In the present project (Multidomain Intervention to preveNt Disability in ElDers, MINDED), we propose to conduct a pilot study aimed at estimating the effects of a multidomain person-tailored preventive intervention (based on physical activity, cognitive training, and nutritional modifications) on frailty status, physical performance, cognitive function, nutritional status, health-related quality of life, and use of health care services. In addition, we will perform cost-effectiveness analyses of the proposed intervention. The project will yield the necessary preliminary data to design a definitive full-scale Phase 3 randomized clinical trial. By providing a conclusive answer about the effectiveness of a multidimensional preventive program in the primary prevention of major health-related outcomes, the results of the full-scale trial will have relevant clinical and public health implications, and will promote the practicing of a truly evidence-based geriatric medicine.

ELIGIBILITY:
Inclusion Criteria:

* Age of 60 years and older;
* Willingness to be randomized to either treatment group;
* Pre-frailty or frailty status according to the phenotype described by Fried and colleagues

Exclusion Criteria:

* Failure to provide informed consent;
* Inability to complete a 400-meter walk test (primary outcome of the study);
* Living in nursing home;
* Living outside of the area of interest, or planning to move out of the area in next 3 years, or planning to leave the area for more than 3 months during the next year;
* Relevant cognitive impairment (defined as a known diagnosis of dementia);
* Severe progressive, degenerative neurologic disease (e.g., multiple sclerosis);
* Severe rheumatologic or orthopaedic diseases (e.g., awaiting joint replacement);
* Terminal illness with life expectancy less than 12 months;
* Severe pulmonary disease (e.g., oxygen therapy or chronic use of steroids);
* Severe cardiac disease (e.g., New York Heart Association Class III or IV heart failure, clinically significant aortic stenosis, history of cardiac arrest, uncontrolled angina);
* Other significant comorbid conditions that would impair the ability to participate in the multidomain intervention (e.g., renal failure on hemodialysis, severe psychiatric disorder, excessive alcohol use). To be noted: persons with depression will not be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-10-16 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01-27 (Actual)

PRIMARY OUTCOMES:
400-meter walk test | 12 months
  Incident inability to complete the 400-meter walk test in the two randomization groups

SECONDARY OUTCOMES:
Participants' adherence/retention to the intervention protocol and control groups | 12 months
  Participants' adherence/retention to the intervention protocol
Intercurrent illnesses rates | 12 months
  Intercurrent illnesses rates in the two randomization groups
Serious fall injuries | 12 months
  Incident fall injuries occurred in the two randomization groups
Hospitalizations and institutionalization rates | 12 months
  Incidence of acute care hospitalizations and nursing home admissions in the two randomization groups
Mortality | 12 months
  Overall mortality rate in the two randomization groups
Health-related quality of life | 12 months
  Modifications of health-related quality of life in the two randomization groups
Body composition modifications | 12 months
  Body composition modifications (assessed using bioimpedance analysis) in the two randomization groups
Modification of Pain | 12 months
  Modification of pain symptoms in the two randomization groups
Fatigue | 12 months
  Modification of the fatigue symptom in the two randomization groups

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Cesari, MD, PhD, Principal Investigator — Inserm UMR1027, Université de Toulouse III Paul Sabatier, Toulouse, France
Locations (1):
- Centre de Rééducation Fonctionnelle "La Roseraie", Montfaucon, France

REFERENCES:
- [Background] Cesari M, Demougeot L, Boccalon H, Guyonnet S, Vellas B, Andrieu S. The Multidomain Intervention to preveNt disability in ElDers (MINDED) project: rationale and study design of a pilot study. Contemp Clin Trials. 2014 May;38(1):145-54. doi: 10.1016/j.cct.2014.04.006. Epub 2014 Apr 24. PMID 24768939